CLINICAL TRIAL: NCT03598621
Title: A Trial to Demonstrate Bioequivalence Between Semaglutide Formulations for the DV3372 Device and the Formulation for the PDS290 Semaglutide Pen-injector
Brief Title: A Research Study to Look at Similarity Between Semaglutide Versions in Different Injection Tools
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9535-4387; U1111-1200-8075 (Other: World Health Organization (WHO)); 2017-003437-29 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1: Semaglutide 0.25 mg (Experimental): Participants will receive a single dose of semaglutide 0.5 mg/mL using DV3372 device and a single dose of semaglutide 1.34 mg/mL using PDS290 device in a cross-over manner at two separate dosing visits. The dosing visits will be separated by a wash-out period of 2-3 weeks.
  Interventions: Drug: Semaglutide, 0.5 mg/mL; Drug: Semaglutide, 1.34 mg/mL; Device: DV3372, 0.5 mg/mL; Device: PDS290
- Cohort 2: Semaglutide 0.5 mg (Experimental): Participants will receive a single dose of semaglutide 1.0 mg/mL using DV3372 device and a single dose of semaglutide 1.34 mg/mL using PDS290 device in a cross-over manner at two separate dosing visits. The dosing visits will be separated by a wash-out period of 2-3 weeks.
  Interventions: Drug: Semaglutide, 1.0 mg/mL; Drug: Semaglutide, 1.34 mg/mL; Device: DV3372, 1.0 mg/mL; Device: PDS290
- Cohort 3: Semaglutide 0.5 mg (Experimental): Participants will receive a single dose of semaglutide 2.0 mg/mL using NovoPen®4 device and a single dose of semaglutide 1.34 mg/mL using PDS290 device in a cross-over manner at two separate dosing visits. The dosing visits will be separated by a wash-out period of 2-3 weeks.
  Interventions: Drug: Semaglutide, 1.34 mg/mL; Drug: Semaglutide, 2.0 mg/mL; Device: PDS290; Device: NovoPen®4

INTERVENTIONS:
Drug: Semaglutide, 0.5 mg/mL — A single dose will be administered subcutaneously (s.c.; under the skin) in the morning after an overnight fast of at least 8 hours.
  Arms: Cohort 1: Semaglutide 0.25 mg
Drug: Semaglutide, 1.0 mg/mL — A single dose will be administered s.c. in the morning after an overnight fast of at least 8 hours.
  Arms: Cohort 2: Semaglutide 0.5 mg
Drug: Semaglutide, 1.34 mg/mL — A single dose will be administered s.c. in the morning after an overnight fast of at least 8 hours.
Drug: Semaglutide, 2.0 mg/mL — A single dose will be administered s.c. in the morning after an overnight fast of at least 8 hours.
  Arms: Cohort 3: Semaglutide 0.5 mg
Device: DV3372, 0.5 mg/mL — DV3372 device will be used for administration of semaglutide 0.5 mg/mL.
  Arms: Cohort 1: Semaglutide 0.25 mg
Device: DV3372, 1.0 mg/mL — DV3372 device will be used for administration of semaglutide 1.0 mg/mL.
  Arms: Cohort 2: Semaglutide 0.5 mg
Device: PDS290 — PDS290 pen-injector will be used for administration of semaglutide 1.34 mg/mL.
Device: NovoPen®4 — NovoPen®4 will be used for administration of semaglutide 2.0 mg/mL.
  Arms: Cohort 3: Semaglutide 0.5 mg

SUMMARY:
This study will compare four different semaglutide versions and different injection tools. The study aims to show similar levels of semaglutide in the blood using different versions of semaglutide. The researchers also want to look at how well the injection tools work. Participants will get two versions of semaglutide at two separate dosing visits. One of them is a version that doctors already can prescribe and the other will be one of the new versions. Which version participants get first is decided by chance. Participants will get semaglutide as an injection under the skin. The time between injections is 7 to 8 weeks. The study will last for about 16 weeks. Participants will have 27 study visits with the study doctor. For two of the visits, participants will stay at the clinic for 4 days and 3 nights.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index between 20.0 and 29.9 kg/m^2 (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol.
* Use of prescription medicinal products or non-prescription drugs or herbal products, except routine vitamins, topical medication, highly effective contraceptives and occasional use of paracetamol, within 14 days prior to the day of screening.
* Abuse or intake of alcohol, defined as any of the below: a) Known or suspected alcohol abuse within 1 year prior to the day of screening (defined as regular intake of more than 24 g alcohol daily for men and 12 g alcohol daily for women. b) Positive alcohol test at screening.
* Abuse or intake of drugs, defined as any of the below: a) Known or suspected drug/chemical substance abuse within 1 year prior to the day of screening. b) Positive drug of abuse test at screening.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using highly affective contraceptive methods.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
AUC0-last,sema,SD, the area under the plasma semaglutide concentration curve from time 0 until last quantifiable measurement after a single dose subcutaneous semaglutide administration | 0-840 hours (5 weeks)
  Measured in nmol·h/L.
Cmax,sema,SD, the maximum plasma semaglutide concentration after a single dose subcutaneous semaglutide administration | 0-840 hours (5 weeks)
  Measured in nmol/L.

SECONDARY OUTCOMES:
AUC0-∞,sema,SD, the area under the plasma semaglutide concentration curve from time 0 until infinity after a single dose subcutaneous semaglutide administration | 0-840 hours (5 weeks)
  Measured in nmol·h/L.
tmax,sema,SD, time to Cmax,sema,SD of semaglutide | 0-840 hours (5 weeks)
  Measured in hours.
t½,sema,SD, terminal elimination half-life of semaglutide | 0-840 hours (5 weeks)
  Measured in hours.
Cl/F,sema,SD, total apparent clearance of semaglutide | 0-840 hours (5 weeks)
  Measured in L/h.
Vz/F,sema,SD, apparent volume of distribution of semaglutide | 0-840 hours (5 weeks)
  Measured in L.
Number of site-initiated technical complaints with or without co-reported adverse events: DV3372 device, 0.5 mg/mL versus PDS290 semaglutide pen-injector, 1.34 mg/mL | Week 0-5 in both treatment period 1 and 2
  Count of technical complaints.
Number of site-initiated technical complaints with or without co-reported adverse events: DV3372 device, 1.0 mg/mL versus PDS290 semaglutide pen-injector, 1.34 mg/mL | Week 0-5 in both treatment period 1 and 2
  Count of technical complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Neuss

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com